CLINICAL TRIAL: NCT01899248
Title: The Effect of Inhalation Agent on the QTc Interval During Liver Transplantation: Sub Study (NCT01886664)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YSJeon_liver transplantation
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sevoflurane: Performing liver transplantation under general anesthesia using sevoflurane
  Interventions: Drug: Sevoflurane
- Desflurane: Performing liver transplantation under general anesthesia using desflurane
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane
  Groups: Sevoflurane
Drug: Desflurane
  Groups: Desflurane

SUMMARY:
The purpose of this study is to assess the effects of inhalation agent on corrected QT interval duration during liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* elective liver transplantation

Exclusion Criteria:

* age < 18, age > 65
* patient refusal
* re-transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who were enrolled prospectively in study (ClinicalTrials.gov Identifier NCT01886664)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
corrected QT interval (QTc interval) | up to postoperative day 1 after surgery
  up to 10 minutes after tracheal intubation, up to 60 minutes after reperfusion, at 10 minutes after hepatectomy, at 10 minutes after biliary anastomosis, at skin closure, at the arrival on ICU, on postoperative day 1.

SECONDARY OUTCOMES:
proportion of patients whose QTc interval is more than 450 ms for men and 470 ms for women | up to postoperative day 1 after surgery
proportion of patients who have more than 500 ms of QTc interval | up to postoperative day 1 after surgery
Tp-e interval | up to postoperative day 1 after surgery
  up to 10 minutes after tracheal intubation, up to 60 minutes after reperfusion, at 10 minutes after hepatectomy, at 10 minutes after biliary anastomosis, at skin closure, at the arrival on ICU, on postoperative day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea